CLINICAL TRIAL: NCT01920542
Title: Renal Effects of Dexmedetomidine During Pediatric Cardiac Surgery: a Randomized Placebo-controlled Study
Brief Title: Dexmedetomidine on Pediatric Heart Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GCIRB2013-163
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Acute Renal Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no dexmedetomidine (Experimental): no administration of dexmedetomidine
  Interventions: Drug: no dexmedetomidine
- dexmedetomidine (Active Comparator): administration of 0.5ug/kg dexmedetomidine for 10 min and infusion of 0.5ug/kg/h of dexmedetomidine until weaning of cardiopulmonary bypass
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — administration of dexmedetomidine on dexemedetomidine group
  Other Names: administration of dexmedetomidine
  Arms: dexmedetomidine
Drug: no dexmedetomidine — no administration of dexmedetomidine on control group
  Other Names: no administration of dexmedetomidine
  Arms: no dexmedetomidine

SUMMARY:
we hypothized dexmedetomidine could reduce the reduction of renal function after cardiopulmonary bypass weaning in pediatric patients

DETAILED DESCRIPTION:
dexmedetomidine, a2-adrenoreceptor agonist has been used for sedation or hemodynamic stability for operative procedure. It had been already reported that dexmedetomidine reduce the impairment of renal functon after cardiac operation in adult. we hypothized dexmedetomidine could reduce the reduction of renal function after cardiopulmonary bypass weaning in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* 1-6yr pediatric cardiac patients

Exclusion Criteria:

* previous renal dysfunction

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
renal function | from anesthetic induction up to postoperative 2h
  at immediate after anesthetic induction (baseline), after weaning of cardiopulmonary bypass, 2h after end of operationCPB, sodium and creatinine in the urine and serum, N-acetyl-b-glucosaminidase (NAG)and albumin in only urine could be studied

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, M.D., Ph.D, Study Director — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Cneter, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided